CLINICAL TRIAL: NCT06962540
Title: Understanding Individual Listening Strategies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00221736
Record Dates: First submitted 2024-12-02; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Speech Recognition; Hearing Aids
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Participants will listen to hearing aids programmed specifically for their listening strategies or to ones programmed with typical clinical settings first, then switch strategies.
Who Masked: Participant
Masking Description: Participants will not know when they are listening to a hearing aid that is programmed with general or customizable settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Customized to match listening strategy First (Active Comparator): Participants in this arm will listen to hearing aid settings programmed to match their listening strategy first, then the general setting
  Interventions: Device: Hearing aid with settings customized to match their individual listening strategy; Device: Hearing Aid with settings based on audiogram alone
- Not customized to match listening strategy First (Active Comparator): Participants will listen to hearing aid settings based only on their pure-tone thresholds first (general hearing aid settings), then ones programmed to match their listening strategies.
  Interventions: Device: Hearing aid with settings customized to match their individual listening strategy; Device: Hearing Aid with settings based on audiogram alone

INTERVENTIONS:
Device: Hearing aid with settings customized to match their individual listening strategy — Behind-the-ear hearing aids that have been programmed based on the participant's individual listening strategy and hearing loss.
  Other Names: Customized Hearing Aid Settings
Device: Hearing Aid with settings based on audiogram alone — Behind-the-ear hearing aids that have been programmed based on their hearing loss and typical clinical settings.
  Other Names: General Hearing Aid Settings

SUMMARY:
The goal of this clinical trial is to learn if hearing aid settings that are customized to individual listening strategies result in better speech understanding than non-customized hearing aid settings. The main question it aims to answer is:

Do customized hearing aid settings result in better speech understanding?

Researchers will compare hearing aid settings that match individual listening strategy to a general setting.

Participants will:

Wear hearing aids for a 2-hour visit to our laboratory. Listen to some sentences in noise and repeat the sentences they hear, with two different hearing aid settings Listen to some sentences in noise and rate how understandable they think those sentences are, with two different hearing aid settings

DETAILED DESCRIPTION:
Participants will complete standard clinical hearing evaluations and a listening profile test to evaluate their individual listening strategy. Hearing aids will then be programmed either based on their clinical hearing evaluations alone using typical hearing aid settings or based on their hearing test with settings further adjusted to account for their individual listening strategies.

ELIGIBILITY:
Inclusion Criteria:

* Sensorineural hearing loss

Exclusion Criteria:

* Montreal Cognitive Assessment < 23 points

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Speech recognition | Outcome measure is collected during the intervention, a two hour visit to the lab where they are wearing the hearing aids
  Participants listen to and repeat sentences, they are scored based on the % correct of keywords they accurately repeat.

SECONDARY OUTCOMES:
Speech Spatial Quality | Outcome measure is collected during the intervention, a two hour visit to the lab where they are wearing the hearing aids
  Rate perceived intelligibility and quality on a scale of 0 to 10 with 10 generally being better

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Souza, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No